CLINICAL TRIAL: NCT04594031
Title: A Phase I Multicenter Study of Hematopoietic Stem Cell Transplant of ECT-001-Expanded Cord Blood With a Reduced Toxicity Conditioning Regimen in Patients With Severe Sickle Cell Disease
Brief Title: US Phase I Study of ECT-001-CB in Patients With Sickle-Cell Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Preference given to gene therapy approaches by the SCD research community and patients' associations
Sponsor: ExCellThera inc. (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT-001.CB.005
Record Dates: First submitted 2020-09-28; First posted 2020-10-20 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Sickle Cell Disease; Umbilical Cord Blood; Hematopoietic Cell Proliferation
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ECT-001-CB (Experimental): * An Umbilical Cord Blood for transplant will undergo CD34+ selection and expansion. The CD34- fraction is infused on Day +1 post-transplant.
  * Patients will receive standard supportive care and GVHD prophylaxis
  Interventions: Biological: ECT-001-CB (UM171-Expanded Cord Blood Transplant)

INTERVENTIONS:
Biological: ECT-001-CB (UM171-Expanded Cord Blood Transplant) — Single ECT-001-CB transplant (CD34+: 2 to 5.75x10E5/kg, CD3+ >1x10E6/kg)

SUMMARY:
The application of experimental hematopoietic cell transplantation (HCT) therapy in sickle-cell disease (SCD) must strike a balance between the underlying disease severity and the possibility of a direct benefit of the treatment, particularly in pediatric populations. Clinical studies in adults with SCD have focused on interventions that prolong survival and improve the quality of life. Unlike children, adults with SCD are much more likely to have a debilitating complication. As a result, the risk/benefit ratio of HCT is very favorable in adults, particularly if an approach to HCT that defines an acceptable level of toxicity can be established.

Whereas hematopoietic stem cell transplantation (HSCT) remains the only curative treatment currently available for patients with SCD, the morbidity, the frequent irreversible damage in target organs and the mortality reported in the natural course of patients with severe SCD are strong incentives to perform HSCTs in younger age groups. For those who lack a matched related donor, CB transplant is an appealing option, but despite been less problematic, CB accessibility related to cell dose of appropriately matched cord blood unit (CBU) remains a significant issue. Through a 7-day culture process of a CBU's hematopoietic stem cell HSCs with the UM171 compound, the total cell dose is increased mitigating this limitation.

UM171-CB expansion (ECT-001-CB) allows a greater CB accessibility, the selection of better matched cords that might translate into favourable clinical outcomes as reported in previous trials, including a lower risk of graft-versus-host disease. After CB selection and ex-vivo expansion, ECT-001-CB transplant will follow a myeloablative reduced-toxicity conditioning regimen consisting of rATG, busulfan and fludarabine with doses of all agents optimized to the individual using model-based dosing and will be followed by standard supportive care and GVHD prophylaxis consisting of tacrolimus and MMF.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 5-30 years of age.
2. Have a diagnosis of SCD, with either βS/βS, βS/β0, βS/β+ or βS/βC genotype and followed at a center of excellence for SCD with at least 2 years of detailed past medical records available.
3. Have severe disease i.e. have experienced one or more of the following SCD related events, in spite of appropriate supportive care measures (e.g. pain management, penicillin prophylaxis):

   1. Recurrent severe vaso-occlusive crisis (VOC) (≥2 episodes/year in the prior 2 years): an episode of pain lasting >2 hours severe enough to require care at a medical facility. Note that priapism that lasts >2 hours and requires care at a medical facility is also considered a VOC. To meet this criterion, subjects must have either experienced hydroxyurea failure at any point in the past (defined as >1 VOC or ≥1 acute chest syndrome (ACS) after taking hydroxyurea for ≥3 months) or must have intolerance to hydroxyurea (defined as inability to be maintained on an adequate dose of hydroxyurea due to marrow suppression or severe drug-induced toxicity [e.g. gastrointestinal distress, fatigue]).
   2. ACS (≥2 total episodes in the prior 2 years, with at least one episode in the past year), defined as an acute event with pneumonia-like symptoms, hypoxemia and the presence of a new pulmonary infiltrate. To meet this criterion, subjects must have either experienced hydroxyurea failure or have intolerance to hydroxyurea, as defined above.
   3. History of an overt stroke, defined as a sudden onset neurologic deficit lasting more than 24 hours that is accompanied by cerebral MRI changes.
   4. patients on chronic transfusions are eligible, provided medical records documenting any of the above severity criteria are available prior to starting the transfusion program.
4. Availability of 1 CB unit ≥ 6/8 HLA match (when A, B, C and DRB1 are performed at the allelic level resolution) with of at least CD34+ cell count 1.5 x 105/kg and total nucleated cells (TNC) 1.5 x 107/kg (pre-freeze)
5. Have adequate organ function to undergo a myeloablative (reduced toxicity conditioning) HSCT.
6. Have a Lansky/Karnofsky performance status of ≥ 80.
7. An appropriate and willing HLA-matched sibling donor is not available.

Exclusion Criteria:

1. Prior HSCT or gene-therapy.
2. Positive for presence of HIV-1 or HIV-2, hepatitis B virus (HBV), or hepatitis C virus (HCV). (Note that patients who have been vaccinated against hepatitis B [hepatitis B surface antibody (HBsAb)-positive] or patients with positive hepatitis B core and/or hepatitis B-e antibodies are also eligible provided viral load is negative by quantitative polymerase chain reaction (qPCR). Patients who are positive for anti-hepatitis C antibody are eligible as long as they have a negative HCV viral load by qPCR). Positive serology for human T-lymphotropic virus-1 (HTLV-1), syphilis (rapid plasma reagin (RPR)), toxoplasmosis.
3. Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by PI.
4. A white blood cell count <2 × 10e9/L, and/or platelet count <50 × 10e9/L.
5. Any prior or current malignancy or myeloproliferative or a significant coagulation or immunodeficiency disorder.
6. Advanced liver disease, defined as:

   1. Persistent aspartate transaminase, alanine transaminase, or direct bilirubin value >5 times the upper limit of normal (ULN); or
   2. Cirrhosis or bridging fibrosis; or
   3. Baseline prothrombin time or partial thromboplastin time > 1.5 x ULN; or
   4. in chronically transfused patients a liver iron concentration (LIC) of ≥ 15 mg/g on T2* Magnetic Resonance Imaging [MRI] of liver.
7. Left ventricular ejection fraction (LVEF) <45% and for patients on chronic transfusions a cardiac T2* < 10 ms by MRI.
8. Baseline estimated glomerular filtration rate < 60 mL/min/1.73 m2.
9. Baseline oxygen saturation < 85% without supplemental oxygen (excluding periods of SCD crisis or infection).
10. Diffusion capacity of carbon monoxide (DLCO) <50% of predicted (corrected for hemoglobin and/or alveolar volume).
11. Any contraindication to general anaesthesia.
12. Participation in another clinical study with an investigational drug within 30 days of Screening.
13. Diagnosis of a significant psychiatric disorder as deemed as the PI that could seriously impede the subject's ability to participate in the study.
14. Pregnancy or breastfeeding in a postpartum female or absence of adequate contraception for fertile patients. Females of child bearing potential are required to use effective contraception from enrollment through at least 6 months after drug product infusion. Male patients are required to use effective contraception from enrollment through at least 6 months after drug product infusion.
15. An assessment by the PI that the subject would not comply with the study procedures outlined in the protocol.
16. Any abnormal condition or laboratory result that is considered by the PI capable of altering patient condition or study outcome.

Note: should a patient be out of range for any numerical exclusion criteria, the PI is allowed to repeat the dosage once during the screening period to definitely determine eligibility

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate feasibility of finding a suitable ECT-001-CB graft for transplantation in the context of SCD. | Up to 24-months
  Calculate the proportion of recruited SCD patients for whom a suitable CBU (i.e., ≥ 6/8 human leukocyte antigen (HLA) with an appropriate cell dose) is identified.
Evaluate feasibility of a successfully performing ECT-001-CB transplantation in the context of SCD. | During accrual (up to 24-months)
  Calculate the percentage of selected grafts that will be successfully expanded and transplanted with absence of technical hurdles
Evaluate the Safety of ECT-001-CB by evaluating tri-lineage hematopoietic reconstitution | Up to 12-Months
  Measure the time required to achieve neutrophil and platelet engraftment
Evaluate the Safety of ECT-001-CB by calculating incidence of acute and chronic GvHD | Up to 12-Months
  Calculate incidence of Acute GVHD and Chronic GVHD as per NIH criteria
Evaluate the Safety of ECT-001-CB by evaluating adverse events | Up to 12-Months
  Calculate the Incidence of Adverse Events from the beginning of the conditioning regimen up to 12 months after ECT-001-CB transplant
Evaluate the Safety of ECT-001-CB by evaluating incidence of transplant related mortality (TRM) | Up to 12-Months
  Calculate incidence of any mortality related to the investigational product until the end of evaluation period.
Evaluate the Safety of ECT-001-CB by incidence of graft failure | Up to 100 days
  Calculate the incidence of primary and late graft failure

SECONDARY OUTCOMES:
Determine the pharmacologic effect of ECT-001-CB by evaluating donor chimerism | Up to 12-Months post treatment
  The percentage of hematopoietic chimerism, based on DNA polymorphisms, will be measured and compared to baseline.
Determine the pharmacologic effect of ECT-001-CB by measuring sickle hemoglobin (HbS) in peripheral blood. | Up to 12-Months post treatment
  The concentration of the Sickle Hemoglobin (HbS) will be compared to baseline.
Evaluate impact of ECT-001-CB on SCD-related events during the study period. | Up to 12-Months post treatment
  The incidence of SCD-related adverse events will be compared to internal controls

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — ExCellThera inc.
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Palo Alto, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No